CLINICAL TRIAL: NCT05496491
Title: Neoadjuvant Chemoradiotherapy and Consolidation Chemotherapy for Rectal Cancer: A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Perivoliotis Konstantinos, Perivoliotis Konstantinos, Principal Investigator, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCRC
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Rectal Neoplasms
Keywords: rectal; cancer; neoadjuvant; radiotherapy; chemotherapy; mesorectal; excision
MeSH Terms: conditions — Rectal Neoplasms; Neoplasms | interventions — Neoadjuvant Therapy; Chemotherapy, Adjuvant; Consolidation Chemotherapy

STUDY DESIGN:
Intervention Model Description: The study will employ a prospective, parallel randomized-controlled design
Masking Description: There will be no blindness at the level of the patient, the treating physicians (surgeon, oncologist, radiotherapist) and the researcher who will record the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant Chemoradiotherapy and Consolidation Chemotherapy (Experimental): The experimental group will receive the standard 5-week neoadjuvant chemoradiotherapy (CRT). Thereafter, all patients will commence consolidation chemotherapy. At the 6th week after the end of CRT, patients will undergo MRI re-staging: In case of non-response (mrTRG 5) they will be submitted immediately to surgery, and, subsequently, excluded from the trial.
  In case of response (mrTRG 2-4) they will receive consolidation chemotherapy for the whole waiting period between the end of CRT and surgery - 12 weeks.
  Interventions: Radiation: Neoadjuvant Chemoradiotherapy; Drug: Consolidation Chemotherapy
- Neoadjuvant Chemoradiotherapy and Adjuvant Chemotherapy (Active Comparator): The control group will receive the standard 5-week neoadjuvant chemoradiotherapy regimen. Six weeks after completion the patient will be re-staged with rectal MRI and depending on the response will be operated (TME): immediately in case of non-response (mrTRG 5) or after an additional 6-week delay (overall 12 weeks after the end of chemoradiotherapy) in case of partial response (mrTRG 2-4). Adjuvant chemotherapy will be, also, administered.
  Interventions: Radiation: Neoadjuvant Chemoradiotherapy; Drug: Adjuvant Chemotherapy

INTERVENTIONS:
Radiation: Neoadjuvant Chemoradiotherapy — 5-week neoadjuvant radiotherapy regimen (28 x 1.8 Gy) combined with Capecitabine (bid 800 mg/m2, twice daily, on days 1-33-38)
  Other Names: nCRT
Drug: Adjuvant Chemotherapy — 8 cycles of CAPOX (Capecitabine bid 1000 mg/m2, twice daily, day 1-14, every 3 weeks and Oxaliplatin 130 mg/m2, day 1, every 3 weeks) or alternatively, 12 cycles of folinate, fluorouracil and oxaliplatin (FOLFOX)
  Other Names: AC
  Arms: Neoadjuvant Chemoradiotherapy and Adjuvant Chemotherapy
Drug: Consolidation Chemotherapy — CAPOX (Capecitabine bid1000 mg/m2 and Oxaliplatin 130 mg/m2, day 1, every 3 weeks) or alternatively FOLFOX
  Other Names: CC
  Arms: Neoadjuvant Chemoradiotherapy and Consolidation Chemotherapy

SUMMARY:
The purpose of this protocol is to compare neoadjuvant chemoradiation plus consolidation chemotherapy before surgical resection with the standard neoadjuvant chemoradiation followed by surgical resection and adjuvant chemotherapy in patients with rectal cancer.

DETAILED DESCRIPTION:
Colorectal cancer is the second leading cause of cancer-related deaths worldwide. It is estimated that 10% of cancer mortality is attributed to malignant neoplasms of the colon and rectum. More specifically, in the United States alone, 53,200 colorectal cancer deaths were reported.

The current treatment of choice for locally advanced rectal cancer (Stage II/ III) is the combination of neoadjuvant chemoradiation followed by radical surgical resection based on the principles of total mesorectal excision (TME) after a 8-12 weeks period. Therapy is usually completed with the administration of adjuvant chemotherapy based on oxaliplatin and fluoropyrimidines. This combined approach allowed the reduction of local recurrence at levels around 5%. Despite the impressive results in local control, the same was not confirmed for the long-term, overall survival. Possible explanations to that are: a) the compliance and completion of the treatment schemes during the postoperative period were low and b) there was a delay in the administration of adjuvant chemotherapy; both could lead to subclinical metastatic disease progression.

On the basis of achieving both goals, (i.e., local control through neoadjuvant radiotherapy and metastatic disease control through systemic chemotherapy) the administration of the two therapies in the preoperative period was proposed, in the form of combined or total neoadjuvant therapy.

Additional theoretical benefits of total neoadjuvant therapy is faster defunctioning stoma reversal, as well as, the possibility of a more accurate evaluation of the tumor biological behavior, thus enabling a safer staging for patients who would be candidates for a watch and wait protocol. Furthermore, for patients who will eventually undergo surgery, total neoadjuvant therapy could probably increase R0 resection and sphincter-preservation rates.

However, many researchers question the safety and efficacy of total neoadjuvant therapy. First, the administration of neoadjuvant chemotherapy significantly increases the risk of severe toxicity from cytotoxic agents. At the same time, according to the results of one of the largest prospective randomized trials, the addition of neoadjuvant chemotherapy into the treatment algorithm did not offer any advantage in the pathological response, 5-year overall and disease-free survival rates. Finally, there is considerable heterogeneity in the current literature, most likely reflecting the different schemes used in different trials regarding the radiotherapy regimen, the chemotherapy regimen as well as the sequence of each one in each protocol.

The investigators believe that it is difficult to interpret any differences in results when multiple parameters have been changed in a comparative trial. For this reason when testing the current standard neoadjuvant protocol to the new trend of total neoadjuvant therapy it was decided to keep the same scheme and timing for the experimental group while the only parameter which was different was the use of the classic chemotherapy scheme during the waiting period following chemoradiation and before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed rectal adenocarcinoma
* cT3, cT4, threatened CRM / MRF, EMVI (+), ≥N1
* Multidisciplinary tumor board decision for neoadjuvant treatment
* Tumor distance from the anal verge <15 cm based on endoscopy or magnetic resonance imaging
* Patient 18 to 80 years old
* General health condition status WHO 0-1
* Absence of co-morbidities that may affect treatment
* Neutrophils >1,500 / mm3, platelets >100,000 / mm3, hemoglobin> 10 g / dL, normal creatinine, and creatinine clearance> 50 mL / min
* Signed informed consent of the patient

Exclusion Criteria:

* Distant metastases
* Non-resectable cancer
* Contraindications for the administration of chemotherapy
* Previous pelvic radiotherapy or chemotherapy
* History of inflammatory bowel disorders
* History of angina, acute myocardial infarction or heart failure
* Active sepsis or systemic infection
* Untreated physical and mental disability
* Synchronous malignancy
* Pregnancy or breast-feeding
* Lack of compliance with the protocol process
* Non-granting of signed informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | 3 years postoperatively
  Occurence of Disease Free Survival. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'

SECONDARY OUTCOMES:
Complete Pathological Response | 1 month postoperatively
  Occurence of Complete Pathological Response. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Postoperative Complication | 1 month postoperatively
  Occurence of postoperative complications based on the Clavien Dindo Classification. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Length of Hospital Stay | Maximum time frame 39 days postoperatively
  Postoperative time that the patient can be safely discharged. Measurement unit: days. The patient will be discharged, when it is ensured that is medically safe to be released. In particular, as the exit time of the patient, will be regarded the time that the patient will fulfil the Clinical Discharge Criteria
Readmission | 1 month postoperatively
  Occurence of postoperative readmission. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Negative Resection Margin | 1 month postoperatively
  Occurence of Negative Resection Margin. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Overall Survival | 3 years postoperatively
  Occurence of Overall Survival. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Chemotherapy Toxicity | 3 years postoperatively
  Occurence of Chemotherapy Toxicity. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Local Recurrence | 3 years postoperatively
  Occurence of Local Recurrence. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Treatment Compliance | 3 years postoperatively
  Occurence of Treatment Compliance. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Perivoliotis, MD, Principal Investigator — University Hospital of Larissa; George Tzovaras, Prof, Study Director — University Hospital of Larissa
Locations (1):
- Department of Surgery, University Hospital of Larissa, Larissa, Greece

IPD SHARING:
Plan to Share IPD: No
No plan to share individual patient data

REFERENCES:
- [Background] Liu S, Jiang T, Xiao L, Yang S, Liu Q, Gao Y, Chen G, Xiao W. Total Neoadjuvant Therapy (TNT) versus Standard Neoadjuvant Chemoradiotherapy for Locally Advanced Rectal Cancer: A Systematic Review and Meta-Analysis. Oncologist. 2021 Sep;26(9):e1555-e1566. doi: 10.1002/onco.13824. Epub 2021 Jun 7. PMID 33987952
- [Background] Kasi A, Abbasi S, Handa S, Al-Rajabi R, Saeed A, Baranda J, Sun W. Total Neoadjuvant Therapy vs Standard Therapy in Locally Advanced Rectal Cancer: A Systematic Review and Meta-analysis. JAMA Netw Open. 2020 Dec 1;3(12):e2030097. doi: 10.1001/jamanetworkopen.2020.30097. PMID 33326026
- [Background] Sutera P, Solomina J, Wegner RE, Abel S, Monga D, Finley G, McCormick J, Kirichenko AV. Post-Operative Morbidity and Mortality Following Total Neoadjuvant Therapy Versus Conventional Neoadjuvant Chemoradiotherapy in Locally Advanced Rectal Cancer. J Gastrointest Cancer. 2021 Sep;52(3):976-982. doi: 10.1007/s12029-020-00401-3. PMID 32936391
- [Background] Chang H, Jiang W, Ye WJ, Tao YL, Wang QX, Xiao WW, Gao YH. Is long interval from neoadjuvant chemoradiotherapy to surgery optimal for rectal cancer in the era of intensity-modulated radiotherapy?: a prospective observational study. Onco Targets Ther. 2018 Sep 21;11:6129-6138. doi: 10.2147/OTT.S169985. eCollection 2018. PMID 30288048
- [Background] Bahadoer RR, Dijkstra EA, van Etten B, Marijnen CAM, Putter H, Kranenbarg EM, Roodvoets AGH, Nagtegaal ID, Beets-Tan RGH, Blomqvist LK, Fokstuen T, Ten Tije AJ, Capdevila J, Hendriks MP, Edhemovic I, Cervantes A, Nilsson PJ, Glimelius B, van de Velde CJH, Hospers GAP; RAPIDO collaborative investigators. Short-course radiotherapy followed by chemotherapy before total mesorectal excision (TME) versus preoperative chemoradiotherapy, TME, and optional adjuvant chemotherapy in locally advanced rectal cancer (RAPIDO): a randomised, open-label, phase 3 trial. Lancet Oncol. 2021 Jan;22(1):29-42. doi: 10.1016/S1470-2045(20)30555-6. Epub 2020 Dec 7. PMID 33301740
- [Background] Giunta EF, Bregni G, Pretta A, Deleporte A, Liberale G, Bali AM, Moretti L, Troiani T, Ciardiello F, Hendlisz A, Sclafani F. Total neoadjuvant therapy for rectal cancer: Making sense of the results from the RAPIDO and PRODIGE 23 trials. Cancer Treat Rev. 2021 May;96:102177. doi: 10.1016/j.ctrv.2021.102177. Epub 2021 Mar 16. PMID 33798955
- [Background] Shi DD, Mamon HJ. Playing With Dynamite? A Cautious Assessment of TNT. J Clin Oncol. 2021 Jan 10;39(2):103-106. doi: 10.1200/JCO.20.02199. Epub 2020 Oct 14. No abstract available. PMID 33052753
- [Background] Ludmir EB, Palta M, Willett CG, Czito BG. Total neoadjuvant therapy for rectal cancer: An emerging option. Cancer. 2017 May 1;123(9):1497-1506. doi: 10.1002/cncr.30600. Epub 2017 Mar 10. PMID 28295220
- [Background] Petrelli F, Trevisan F, Cabiddu M, Sgroi G, Bruschieri L, Rausa E, Ghidini M, Turati L. Total Neoadjuvant Therapy in Rectal Cancer: A Systematic Review and Meta-analysis of Treatment Outcomes. Ann Surg. 2020 Mar;271(3):440-448. doi: 10.1097/SLA.0000000000003471. PMID 31318794
- [Background] Conroy T, Bosset JF, Etienne PL, Rio E, Francois E, Mesgouez-Nebout N, Vendrely V, Artignan X, Bouche O, Gargot D, Boige V, Bonichon-Lamichhane N, Louvet C, Morand C, de la Fouchardiere C, Lamfichekh N, Juzyna B, Jouffroy-Zeller C, Rullier E, Marchal F, Gourgou S, Castan F, Borg C; Unicancer Gastrointestinal Group and Partenariat de Recherche en Oncologie Digestive (PRODIGE) Group. Neoadjuvant chemotherapy with FOLFIRINOX and preoperative chemoradiotherapy for patients with locally advanced rectal cancer (UNICANCER-PRODIGE 23): a multicentre, randomised, open-label, phase 3 trial. Lancet Oncol. 2021 May;22(5):702-715. doi: 10.1016/S1470-2045(21)00079-6. Epub 2021 Apr 13. PMID 33862000
- [Background] Jimenez-Rodriguez RM, Quezada-Diaz F, Hameed I, Kalabin A, Patil S, Smith JJ, Garcia-Aguilar J. Organ Preservation in Patients with Rectal Cancer Treated with Total Neoadjuvant Therapy. Dis Colon Rectum. 2021 Dec 1;64(12):1463-1470. doi: 10.1097/DCR.0000000000002122. PMID 34508014
- [Background] Bauer PS, Chapman WC Jr, Atallah C, Makhdoom BA, Damle A, Smith RK, Wise PE, Glasgow SC, Silviera ML, Hunt SR, Mutch MG. Perioperative Complications After Proctectomy for Rectal Cancer: Does Neoadjuvant Regimen Matter? Ann Surg. 2022 Feb 1;275(2):e428-e432. doi: 10.1097/SLA.0000000000003885. PMID 32209914
- [Background] Sclafani F, Corro C, Koessler T. Debating Pros and Cons of Total Neoadjuvant Therapy in Rectal Cancer. Cancers (Basel). 2021 Dec 18;13(24):6361. doi: 10.3390/cancers13246361. PMID 34944980
- [Background] Fernandez-Martos C, Garcia-Albeniz X, Pericay C, Maurel J, Aparicio J, Montagut C, Safont MJ, Salud A, Vera R, Massuti B, Escudero P, Alonso V, Bosch C, Martin M, Minsky BD. Chemoradiation, surgery and adjuvant chemotherapy versus induction chemotherapy followed by chemoradiation and surgery: long-term results of the Spanish GCR-3 phase II randomized trialdagger. Ann Oncol. 2015 Aug;26(8):1722-8. doi: 10.1093/annonc/mdv223. Epub 2015 May 8. PMID 25957330
- [Background] Marco MR, Zhou L, Patil S, Marcet JE, Varma MG, Oommen S, Cataldo PA, Hunt SR, Kumar A, Herzig DO, Fichera A, Polite BN, Hyman NH, Ternent CA, Stamos MJ, Pigazzi A, Dietz D, Yakunina Y, Pelossof R, Garcia-Aguilar J; Timing of Rectal Cancer Response to Chemoradiation Consortium. Consolidation mFOLFOX6 Chemotherapy After Chemoradiotherapy Improves Survival in Patients With Locally Advanced Rectal Cancer: Final Results of a Multicenter Phase II Trial. Dis Colon Rectum. 2018 Oct;61(10):1146-1155. doi: 10.1097/DCR.0000000000001207. PMID 30192323
- [Background] Fang Y, Sheng C, Ding F, Zhao W, Guan G, Liu X. Adding Consolidation Capecitabine to Neoadjuvant Chemoradiotherapy for Locally Advanced Rectal Cancer: A Propensity-Matched Comparative Study. Front Surg. 2022 Jan 27;8:770767. doi: 10.3389/fsurg.2021.770767. eCollection 2021. PMID 35155545
- [Background] Chakrabarti D, Rajan S, Akhtar N, Qayoom S, Gupta S, Verma M, Srivastava K, Kumar V, Bhatt MLB, Gupta R. Short-course radiotherapy with consolidation chemotherapy versus conventionally fractionated long-course chemoradiotherapy for locally advanced rectal cancer: randomized clinical trial. Br J Surg. 2021 May 27;108(5):511-520. doi: 10.1093/bjs/znab020. PMID 33724296
- [Background] Wu H, Fan C, Fang C, Huang L, Li Y, Zhou Z. Preoperative short-course radiotherapy followed by consolidation chemotherapy for treatment with locally advanced rectal cancer: a meta-analysis. Radiat Oncol. 2022 Jan 24;17(1):14. doi: 10.1186/s13014-021-01974-4. PMID 35073940
- [Background] Seo N, Kim H, Cho MS, Lim JS. Response Assessment with MRI after Chemoradiotherapy in Rectal Cancer: Current Evidences. Korean J Radiol. 2019 Jul;20(7):1003-1018. doi: 10.3348/kjr.2018.0611. PMID 31270972
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Chung F, Chan VW, Ong D. A post-anesthetic discharge scoring system for home readiness after ambulatory surgery. J Clin Anesth. 1995 Sep;7(6):500-6. doi: 10.1016/0952-8180(95)00130-a. PMID 8534468
- [Background] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190

DOCUMENTS (2):
  • Study Protocol (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT05496491/Prot_000.pdf
  • Informed Consent Form (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT05496491/ICF_001.pdf